CLINICAL TRIAL: NCT04966572
Title: Short Term Efficiency of Presurgical Vacuum Formed Nasoalveolar Molding Aligners in Infants With Bilateral Cleft Lip and Palate Compared With Conventional Grayson Acrylic Formed Nasoalveolar Molding Appliances: A Randomized Clinical Trial
Brief Title: Short Term Efficiency of Presurgical Vacuum Formed Nasoalveolar Molding Aligners in Infants With Bilateral Cleft Lip and Palate Compared With Grayson Acrylic Formed Nasoalveolar Molding Appliances.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khadega Ali Al Khateeb, Phd student, faculty of Dentistry, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCLP_ Grayson_ vacuum
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Cleft Lip and Palate; Bilateral Cleft Lip/Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Presurgical vacuum formed nasoalveolar molding aligners group (Experimental): In this group, all patients will receive 1-2 VF-NAM aligners incorporated with palatal screw in addition to taping from day 1 for 4-6 Months with follow-up every 3 weeks
  Interventions: Device: Presurgical vacuum formed nasoalveolar molding aligners
- conventional Grayson acrylic formed nasoalveolar molding appliances group (Experimental): This group will receive conventional Grayson acrylic formed nasoalveolar molding appliances without taping except some cases, with follow up every week for activation.
  Interventions: Device: Conventional Grayson acrylic formed nasoalveolar molding appliances

INTERVENTIONS:
Device: Presurgical vacuum formed nasoalveolar molding aligners — at first visit, the infants will receive this appliance which is a maxillary vacuum plate incorporated with palatal screw, the infant's parents will be instructed to activate the screw and apply horizontal tap which will be placed at the base of nose in order to approximate lip segments and to change tape daily. After that, The infants will be recalled one week after the first visit to add the nasal stents into the appliance.
  Arms: Presurgical vacuum formed nasoalveolar molding aligners group
Device: Conventional Grayson acrylic formed nasoalveolar molding appliances — at first visit, the infants will receive this appliance which is a maxillary acrylic plate without adding taping, the infants will be recalled bi weekly for activating the appliance.
  When the cleft alveolar gap is reduced to 6mm or less, a pair of nasal stents will be added to mold the nasal cartilage. the infants will be followed up for 4-6 months.
  Arms: conventional Grayson acrylic formed nasoalveolar molding appliances group

SUMMARY:
Newborns with bilateral cleft lip/ palate will be treated pre-surgically by either presurgical vacuum-formed nasoalveolar molding aligners VF (NAM) or conventional Grayson acrylic formed nasoalveolar molding appliances in order to evaluate their effect on the maxillary arch.

DETAILED DESCRIPTION:
The aim of this trial is to evaluate and compare the short-term effect of VF (NAM) aligners with conventional Grayson appliances at 2 stages T1 (Before NAM therapy), and T2 (After NAM therapy) as regards maxillary arch changes.

Newborns with Bilateral cleft lip/ palate will be allocated randomly into two groups: the first group will receive presurgical vacuum-formed nasoalveolar molding aligners while the second group will receive conventional Grayson acrylic formed nasoalveolar molding appliances. The follow-up period will be 4-6 months till surgical lip closure. The changes in the maxillary arch will be assessed by digital maxillary models.

ELIGIBILITY:
Inclusion Criteria:

* Non-syndromic Infants with complete BCLP infants
* Infants less than 1 month of age
* Males and females.
* Infants with displaced premaxilla
* Patients whose parents provided written consent for the study.

Exclusion Criteria:

* Patients above 1 month of age
* Syndromic and systemically ill infants.
* Patients with unilateral cleft lip and palate.
* Incomplete Cleft lip.
* Medically compromised patients
* Patient's/guardians who will be unwilling to go through the PNAM therapy

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the maxillary arch | T1 and T2 (4- 6 months)
  they will be measured in mm by digital models

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Abdu Abdelsayed, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Khateeb KA, Aboulfotouh MH, Abdelsayed F, Mohamed W, Abd-El-Ghafour M. Three-dimensional assessment of maxillary arch changes in infants with bilateral cleft lip and palate using vacuum-formed nasoalveolar molding with active screw versus conventional nasoalveolar molding appliances: a randomized clinical trial. BMC Oral Health. 2025 Aug 19;25(1):1339. doi: 10.1186/s12903-025-06607-w. PMID 40830787